CLINICAL TRIAL: NCT02371538
Title: A Pilot Study of Enteral Donor Human Milk in Young Children With Norovirus Infection of the Gut
Brief Title: Human Breastmilk in Young Children With Norovirus Infection of the Gut
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Mothers' Milk Bank Northeast (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-3363
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Norovirus Infections
Keywords: stem cell transplant; human breastmilk
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor Breastmilk (Experimental): Donated human milk is subjected to pasteurization prior to use. Milk consumption is to be overseen by a Registered Dietician. Oral or enteral milk feeding will begin at 180 ml/day and will be advanced as quickly as tolerated to a goal of 360 ml/day for 6 weeks. If symptoms and stool tests for norovirus do not improve after 6 weeks, milk administration may continue for an additional 6 weeks.
  Interventions: Dietary Supplement: Donor Breastmilk

INTERVENTIONS:
Dietary Supplement: Donor Breastmilk — Donor breastmilk will be obtained from the Mother's Milk Bank of New England.

SUMMARY:
Human Breast milk in young children with Norovirus Infection

DETAILED DESCRIPTION:
The investigators hypothesize that children with clinically significant norovirus infection of the gut who receive enteral human milk will more successfully clear the virus or experience improved symptoms compared to children not receiving human milk.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least two stool samples taken at least 7 days apart that are positive for norovirus
* Child has an underlying disease or has received immunosuppressive medication or chemotherapy such that clearance of norovirus is expected to be impaired.

Exclusion Criteria:

* The presence of other pathogens causing diarrhea that have specific treatments does not preclude enrollment. However, specific treatment should be offered in addition to human milk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07-02 (Actual); Study Completion 2016-07-02 (Actual)

PRIMARY OUTCOMES:
Loose/Unformed/Liquid Stools or Abdominal Cramping | Up to 12 weeks
  Episodes or number of days of loose/unformed/liquid stools or abdominal cramping will be reported.
Norovirus | Up to 12 weeks
  Stool samples will be tested for the presence of norovirus.

CONTACTS AND LOCATIONS:
Overall Officials: Javier El-Bietar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States